CLINICAL TRIAL: NCT02937571
Title: Carfilzomib, Lenalidomide, and Dexamethasone in Newly-Diagnosed Multiple Myeloma: A Clinical and Correlative Phase I/II Dose Escalation Study
Brief Title: High Dose Carfilzomib for Newly Diagnosed Myeloma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Onyx/Amgen (Unknown); Celgene (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15-326
Record Dates: First submitted 2016-10-17; First posted 2016-10-18 (Estimated); Results first posted 2025-11-20 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2024-10

CONDITIONS: Multiple Myeloma
Keywords: Carfilzomib; Lenalidomide; Dexamethasone; 15-326
MeSH Terms: conditions — Multiple Myeloma | interventions — carfilzomib; Lenalidomide; Dexamethasone

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Carfilzomib, Lenalidomide, and Dexamethasone (Experimental): * Cycle 1 ONLY: Carfilzomib 20 mg/m2 per dose, days 1 and 2; Carfilzomib 45 or 56 mg/m2 per dose, days 8, 9, 15, and 16.
  * Cycles 2- up to 12: Carfilzomib 45 or 56 mg/m2 per dose, days 1, 2, 8, 9, 15, and 16
  * Cycles 1- up to 12: Lenalidomide 25 mg/day, days 1-21 every 28 days
  * Cycles 1-4: Dexamethasone 20 mg/dose, days 1, 2, 8, 9, 15, 16, 22, and 23
  * Cycles 5- up to 12: Dexamethasone 10 mg/dose, days 1, 2, 8, 9, 15, 16, 22 and 23
  Interventions: Drug: Carfilzomib; Drug: Lenalidomide; Drug: Dexamethasone

INTERVENTIONS:
Drug: Carfilzomib
Drug: Lenalidomide
Drug: Dexamethasone

SUMMARY:
The purpose of this study is to test whether giving high doses of carfilzomib along with the other drugs (lenalidomide and dexamethasone) is safe and which dose is best tolerated by patients. In addition, the study is designed to test the amount of remaining myeloma cells in the body after treatment with higher carfilzomib doses which is known as minimal residual disease (MRD).

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed patients with histologically confirmed MM based on the following criteria:

  * Clonal plasma cells in the bone marrow
  * Measurable disease within the past 4 weeks defined by any one of the following:
* Serum monoclonal protein ≥ 1.0 g/dL
* Urine monoclonal protein >200 mg/24 hour
* Involved serum immunoglobulin free light chain > 10 mg/dL AND abnormal kappa/lambda ratio
* Evidence of underlying end organ damage and/or myeloma defining event attributed to underlying plasma cell proliferative disorder meeting at least one of the following:

  * Hypercalcemia: serum calcium >0.25 mmol/L (> 1 mg/dL) above upper limit of normal or ≥ 2.75 mmol/L (11 mg/dL)
  * Anemia: hemoglobin value <10 g/dL or > 2 g/dL below lower limit of normal
  * Bone disease: ≥ 1 lytic lesions on skeletal X-ray, CT, or PET-CT. For patients with 1 lytic lesion, bone marrow should demonstrate ≥10% clonal plasma cells
  * Clonal bone marrow plasma cell percentage ≥60%
  * Involved/un-involved serum free light chain ratio ≥100 and involved free light chain >100 mg/L.

    * 1 focal lesion on magnetic resonance imaging study (lesion must be >5 mm) in size
* Creatinine Clearance ≥ 60 ml/min. CrCl can be measured or estimated using Cockcroft-Gault method
* Age ≥ 18 years at the time of signing the informed consent documentation
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* Absolute neutrophil count (ANC) ≥ 1.0 K/uL, hemoglobin ≥ 8 g/dL, and platelet count ≥ 75 K/uL, unless if cytopenias are deemed to be due disease at discretion of clinical investigator. Transfusions and growth factors are permissible.
* Adequate hepatic function, with bilirubin < 1.5 x the ULN, and AST and ALT < 3.0 x ULN.
* All study participants must be able to tolerate one of the following thromboprophylactic strategies: aspirin, low molecular weight heparin or warfarin (coumadin) or alternative anti-coagulant.
* All study participants must be registered into the mandatory eREMS® program, and be willing and able to comply with the requirements of REMS®.
* Females of childbearing potential (FCBP)† must have a negative serum or urine pregnancy test within 10 - 14 days and again within 24 hours prior to prescribing lenalidomide for Cycle 1 (prescriptions must be filled within 7 days) and must either commit to continued abstinence from heterosexual intercourse or begin TWO acceptable methods of birth control, one highly effective method and one additional effective method AT THE SAME TIME, at least 28 days before she starts taking lenalidomide. FCBP must also agree to ongoing pregnancy testing. Men must agree to use a latex condom during sexual contact with a FCBP even if they have had a successful vasectomy.

  * A female of childbearing potential is a sexually mature female who: 1) has not undergone a hysterectomy or bilateral oophorectomy; or 2) has not been naturally postmenopausal for at least 24 consecutive months (i.e., has had menses at any time in the preceding 24 consecutive months).

Exclusion Criteria:

* Patients receiving >1 cycle of prior treatment or concurrent systemic treatment for multiple myeloma.

  * Treatment of hypercalcemia or spinal cord compression or aggressively progressing myeloma with current or prior corticosteroids is permitted
  * Bisphosphonates are permitted
  * Concurrent or prior treatment with corticosteroids for indications other than multiple myeloma is permitted
  * Prior treatment with radiotherapy is permitted
  * Prior treatment for smoldering myeloma is permitted with a washout period of 4 weeks from last dose. Smoldering patients previously treated with carfilzomib are excluded.
  * Patients with measurable disease who received up to one cycle of any therapy within 60 days with a washout period of 4 weeks from last dose (on a trial or outside a trial) are eligible
* Plasma cell leukemia
* POEMS syndrome
* Amyloidosis
* Pregnant or lactating females. Because there is a potential risk for adverse events nursing infants secondary to treatment of the mother with carfilzomib in combination with lenalidomide. These potential risks may also apply to other agents used in this study.
* Uncontrolled hypertension or diabetes
* Active hepatitis B or C infection
* Known or suspected HIV or serologically positive
* Has significant cardiovascular disease with NYHA Class III or IV symptoms, EF<40% or hypertrophic cardiomyopathy, or restrictive cardiomyopathy, or myocardial infarction within 6 months prior to enrollment, or unstable angina, or unstable arrhythmia as determined by history and physical examination. Echocardiogram will be performed during screening evaluation.
* Moderate or severe pulmonary hypertension defined as PASP > 50mm Hg. For those patients were PASP is indeterminate, moderate to severe symptoms of pulmonary hypertension (World Health Organization functional assessment class III or IV) will be used to determine exclusion criteria.
* Has refractory GI disease with refractory nausea/vomiting, inflammatory bowel disease, or bowel resection that would prevent absorption of oral agents
* Uncontrolled intercurrent illness including but not limited to active infection or psychiatric illness/social situations that would compromise compliance with study requirements
* Significant neuropathy ≥Grade 3 or Grade 2 neuropathy with pain at baseline
* Contraindication to any concomitant medication, including antivirals or anticoagulation
* Major surgery within 3 weeks prior to first dose

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2016-10; Primary Completion 2024-10-08 (Actual); Study Completion 2024-10-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Neha Korde, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (6):
- United States (6):
  - Memorial Sloan Kettering Cancer Center, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth, Middletown, New Jersey
  - Memorial Sloan Kettering Bergen, Montvale, New Jersey
  - Memorial Sloan Kettering Cancer Center @ Suffolk, Commack, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — https://www.mskcc.org/

RESULTS

PARTICIPANT FLOW:
Groups:
- Dose Level 1: Carfilzomib 45mg/m2/Dose; Dose Level 2: Carfilzomib 56mg/m2/Dose; MTD: Carfilzomib 56mg/m^2/Dose: * Cycle 1 ONLY: Carfilzomib 20 mg/m2 per dose, days 1 and 2; Carfilzomib 45 or 56 mg/m2 per dose, days 8, 9, 15, and 16.
  * Cycles 2- up to 12: Carfilzomib 45 or 56 mg/m2 per dose, days 1, 2, 8, 9, 15, and 16
  * Cycles 1- up to 12: Lenalidomide 25 mg/day, days 1-21 every 28 days
  * Cycles 1-4: Dexamethasone 20 mg/dose, days 1, 2, 8, 9, 15, 16, 22, and 23
  * Cycles 5- up to 12: Dexamethasone 10 mg/dose, days 1, 2, 8, 9, 15, 16, 22 and 23
  Carfilzomib
  Lenalidomide
  Dexamethasone
Period: Overall Study
Arm/Group | Dose Level 1: Carfilzomib 45mg/m2/Dose | Dose Level 2: Carfilzomib 56mg/m2/Dose | MTD: Carfilzomib 56mg/m^2/Dose
Started | 3 | 3 | 23
Completed | 3 | 3 | 16
Not Completed | 0 | 0 | 7
Not completed — Adverse Event | 0 | 0 | 4
Not completed — Withdrawal by Subject | 0 | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- MTD: Carfilzomib: * Cycle 1 ONLY: Carfilzomib 20 mg/m2 per dose, days 1 and 2; Carfilzomib 45 or 56 mg/m2 per dose, days 8, 9, 15, and 16.
  * Cycles 2- up to 12: Carfilzomib 45 or 56 mg/m2 per dose, days 1, 2, 8, 9, 15, and 16
  * Cycles 1- up to 12: Lenalidomide 25 mg/day, days 1-21 every 28 days
  * Cycles 1-4: Dexamethasone 20 mg/dose, days 1, 2, 8, 9, 15, 16, 22, and 23
  * Cycles 5- up to 12: Dexamethasone 10 mg/dose, days 1, 2, 8, 9, 15, 16, 22 and 23
  Carfilzomib
  Lenalidomide
  Dexamethasone
- Total: Total of all reporting groups
Arm/Group | Dose Level 1: Carfilzomib 45mg/m2/Dose | Dose Level 2: Carfilzomib 56mg/m2/Dose | MTD: Carfilzomib | Total
Number analyzed (Participants) | 3 | 3 | 23 | 29
Age, Continuous [Mean (Full Range); unit: years] | 63 [60 to 66] | 68 [50 to 71] | 60 [43 to 75] | 61 [43 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 10 | 14
  Male | 1 | 1 | 13 | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 2 | 2
  Not Hispanic or Latino | 3 | 3 | 21 | 27
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 3 | 4
  White | 2 | 3 | 16 | 21
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 4 | 4
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 3 | 3 | 23 | 29

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Dose Limiting Toxicity
Description: To find the maximum tolerated dose.A DLT is defined as any of the below toxicities with attribution to one or more of the study drugs that occur during Cycle 1. All AEs should be considered relevant to determining dose-limiting toxicities and to reporting unless the event can clearly be determined to be UNRELATED to the drug. NCI Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 will be utilized for AE reporting.
Time Frame: Cycle 1, up to 28 days
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Level 1: Carfilzomib 45mg/m2/Dose | Dose Level 2: Carfilzomib 56mg/m2/Dose | MTD: Carfilzomib
Number analyzed (Participants) | 3 | 3 | 23
Participants
  Number of participants with DLT | 0 | 0 | 0
  Number of participants without DLT | 3 | 3 | 23

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Dose Level 1: Carfilzomib 45mg/m2/Dose | Dose Level 2: Carfilzomib 56mg/m2/Dose | MTD: Carfilzomib
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/3 | 4/23
Serious Adverse Events (participants affected / at risk) | 0/3 | 1/3 | 15/23
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 23/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dose Level 1: Carfilzomib 45mg/m2/Dose (N=3) | Dose Level 2: Carfilzomib 56mg/m2/Dose (N=3) | MTD: Carfilzomib (N=23)
Chest Pain- Cardiac (Cardiac disorders) | 0 | 0 | 1
Lung Infection (Infections and infestations) | 0 | 0 | 4
Diarrhea (Gastrointestinal disorders) | 0 | 0 | 1
White Blood Cell Decrease (Investigations) | 0 | 0 | 1
Hepatitis Viral (Infections and infestations) | 0 | 0 | 1
Febrile Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1
Upper respiratory Infection (Infections and infestations) | 0 | 0 | 1
Gastrointestinal Perforation (Gastrointestinal disorders) | 0 | 0 | 1
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Platelet count decrease (Investigations) | 0 | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Ejection fraction decreased (Cardiac disorders) | 0 | 0 | 1
Right ventricular dysfunction (Cardiac disorders) | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1
Blood bilirubin increased (Investigations) | 0 | 0 | 1
Acute kidney Injury (Renal and urinary disorders) | 0 | 0 | 1
Thromboembolic Event (Vascular disorders) | 0 | 0 | 2
Constipation (Gastrointestinal disorders) | 0 | 0 | 2
Myocardial infarction (Cardiac disorders) | 0 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1
Rectal Hemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Tooth infection (Infections and infestations) | 0 | 1 | 0
Urinary Retention (Renal and urinary disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dose Level 1: Carfilzomib 45mg/m2/Dose (N=3) | Dose Level 2: Carfilzomib 56mg/m2/Dose (N=3) | MTD: Carfilzomib (N=23)
Activated partial thromboplastin time prolonged (Investigations) | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 1 | 0 | 2
Anemia (Blood and lymphatic system disorders) | 0 | 0 | 12
Anxiety (Psychiatric disorders) | 0 | 1 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 2
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Blood bilirubin increased (Investigations) | 0 | 0 | 1
Cataract (Eye disorders) | 0 | 0 | 2
Constipation (Gastrointestinal disorders) | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 2
Diarrhea (Gastrointestinal disorders) | 0 | 0 | 1
Ejection fraction decreased (Cardiac disorders) | 0 | 0 | 1
Fatigue (General disorders) | 0 | 0 | 2
Fibrinogen decreased (Investigations) | 0 | 0 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 0 | 3
Hyperkalemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 1 | 2
Hyperuricemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypocalcemia (Metabolism and nutrition disorders) | 0 | 1 | 6
Hypokalemia (Metabolism and nutrition disorders) | 1 | 0 | 2
Hyponatremia (Metabolism and nutrition disorders) | 1 | 0 | 4
Hypophosphatemia (Metabolism and nutrition disorders) | 1 | 1 | 11
Lung infection (Infections and infestations) | 0 | 0 | 4
Lymphocyte count decreased (Investigations) | 2 | 1 | 17
Myocardial infarction (Cardiac disorders) | 0 | 0 | 1
Neutrophil count decreased (Investigations) | 0 | 0 | 15
Pain (General disorders) | 0 | 0 | 1
Platelet count decreased (Investigations) | 0 | 1 | 13
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 1 | 6
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 0 | 0 | 1
Skin infection (Infections and infestations) | 2 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 1
Thromboembolic event (Vascular disorders) | 0 | 0 | 2
Tooth infection (Infections and infestations) | 0 | 1 | 0
White blood cell decreased (Investigations) | 0 | 1 | 14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-10-08): https://cdn.clinicaltrials.gov/large-docs/71/NCT02937571/Prot_SAP_000.pdf